CLINICAL TRIAL: NCT00002399
Title: A Multicenter, Randomized, Double-Blind, Phase II Study to Evaluate the Safety, Tolerance and Efficacy of Multiple Doses of SCH 56592 Versus Fluconazole in the Treatment of Oropharyngeal Candidiasis (OPC) in HIV-Positive Patients
Brief Title: A Comparison of SCH 56592 and Fluconazole in the Treatment of Oropharyngeal Candidiasis (OPC) in HIV-Positive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Schering-Plough (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 288A; C96-209; I96-209
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-01

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Fluconazole; Antifungal Agents; Candidiasis; Triazoles
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; AIDS-Related Opportunistic Infections; Candidiasis | interventions — posaconazole; Fluconazole

INTERVENTIONS:
Drug: Posaconazole
Drug: Fluconazole

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of SCH 56592 with that of fluconazole in the treatment of OPC (a fungal infection of the throat) in HIV-positive patients.

DETAILED DESCRIPTION:
This is a randomized, multicenter, double-blind study consisting of 5 arms (4 dose levels of SCH 56592 vs fluconazole) in the treatment of oropharyngeal candidiasis (OPC) in HIV-positive patients.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV seropositivity (by Western blot or other approved confirmatory test) prior to enrollment.
* Pseudomembranous oropharyngeal candidiasis.
* Fungal stain or KOH consistent with Candida species, confirmed by a positive mycologic culture.
* Ability to swallow study medication.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms and conditions are excluded:

* Medical condition requiring use of prohibited drugs.
* Primary HIV seroconversion-related mucosal candidiasis.
* Systemic candidiasis.
* All forms of OPC other than pseudomembranous (unless accompanied by pseudomembranous OPC).
* Documented or suspected fungal esophagitis in patients with symptoms of esophagitis.
* EKG with prolonged QTc interval or clinically-significant abnormalities.

Concurrent Medication:

Excluded:

* Systemic antifungals (IV or oral).
* Topical oral antifungals, e.g., Nystatin, Mycelex, etc.
* Medications known to interact with azoles and that may lead to life-threatening side effects:
* terfenadine, astemizole, cisapride, ebastine, triazolam, midazolam.
* Medications known to lower the serum concentration/efficacy of azole antifungals:
* rifampin, carbamazepine, phenytoin, rifabutin, barbiturates, isoniazid, H2 blockers.
* Cytokines (except erythropoietin), interferon, or lymphocyte replacement therapy unless patient already taking these agents for at least 30 days prior to enrollment.
* Protease inhibitors, starting for the first time, 30 days prior to study enrollment.
* Cytotoxic therapy for cancer.
* Oral or intravenous corticosteroids at supraphysiologic doses (prednisone 10 mg/day or greater; hydrocortisone 40 mg/day or greater; dexamethasone 2 mg/day or greater.

Patients with any of the following prior conditions are excluded:

* Prior enrollment in this study.
* Less than 3 months life expectancy.
* History of hypersensitivity to azole antifungals.
* History of failed therapy with fluconazole 100 mg/day for 2 weeks in the last 3 months.

Prior Medication:

Excluded (wash-outs for medications):

* Systemic antifungals (IV, oral) within 14 days prior to enrollment.
* Topical oral antifungals within 1 day prior to enrollment.
* Oral or intravenous corticosteroids at supraphysiologic doses within 10 days prior to enrollment.
* Astemizole within 10 days prior to enrollment.
* Drugs known to lower the serum concentration/efficacy of azole antifungals within 30 days prior to enrollment.
* Investigational drug (unlicensed new chemical entity) use within 30 days prior to enrollment.

Current known drug abuse, in the opinion of the lead investigator, that would interfere with the subject's participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500

CONTACTS AND LOCATIONS:
Locations (53):
- United States (17):
  - Tucson Veterans Administration Med Ctr, Tucson, Arizona
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Mercy Hosp, Miami, Florida
  - Ponce de Leon Med Ctr, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - Rush Med College / Rush Presbyterian - St Luke's Med Cen, Chicago, Illinois
  - Wishard Hosp, Indianapolis, Indiana
  - Wayne State Univ / Harper Hosp, Detroit, Michigan
  - St Michaels Med Ctr, Newark, New Jersey
  - Duke Univ Med Ctr, Durham, North Carolina
  - Thomas Jefferson Univ / Division of Infectious Disease, Philadelphia, Pennsylvania
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Univ of Texas / Med School at Houston, Houston, Texas
  - Univ of Texas Health Sciences Ctr, San Antonio, Texas
  - Infections Ltd / Physicians Med Ctr, Tacoma, Washington
- Argentina (2):
  - Centro de Micologia / Facultad de Medicina UBA, Buenos Aires
  - Hosp Fernandez, Buenos Aires
- CHU Saint Pierre, Brussels, Belgium
- Canada (3):
  - St Paul's Hosp, Vancouver, British Columbia
  - Victoria Gen Hosp, Halifax, Nova Scotia
  - Montreal Gen Hosp, Montreal, Quebec
- Fundacion Arriaran, Santiago, Chile
- Avenida Lope de Vega Avenue esq/Calle Jose Amado Soler, Ensanche Naco/ Santo Domingo, Dominican Republic
- Faculty of Medicine / Dept of Internal Medicine, Addis Ababa, Ethiopia
- France (8):
  - Hopital Raymond Poincare, Garches
  - Hopital de La Conception, Maseille
  - Hopital Guy de Chauliac Service des Maladies Infectieuses, Montpellier
  - Service des Maladies Infectieuses Hopital de l Archet, Nice
  - Hopital de l Institut Pasteur, Paris
  - Hopital Rothchild, Paris
  - Service des Maladies Infectieuses, Tours
  - Service des Maladies Infectieuses, Villejuif
- Germany (7):
  - Rheinische Friedrich Wilhelms Universitaet Medizinische, Bonn
  - Universitaet Klinik Koln, Cologne
  - Heinrich Heine Universitat, Düsseldorf
  - Allgemeines Krankenhaus St Georg, Hamburg
  - Universitaets Krankenhaus Eppendorf Medizinische Kernklinik, Hamburg
  - Staedtisches Krankenhaus Kiel, Kiel
  - Universitat Munchen / Medizinische Poliklinik, Munich
- Hosp Roosevelt Chief Infectious Diseases Unit, Guatemala City, Guatemala
- Hosp Regional del Seguro Social, San Pedro Sula, Honduras
- Sheba Med Ctr, Tel Litwinsky, Israel
- Hosp de Especialidades Centro Medico La Raza, México, Mexico
- Royal Ctr, Panama City, Panama
- South Africa (3):
  - Daniel Rudolph Malan, Port Elizabeth
  - The Studio, Rosebank
  - Univ of Stellenbosch Med School Depart Med Phys, Tygerberg
- Spain (2):
  - Hosp Clinic, Barcelona
  - Hosp Valle D Hebron, Barcelona
- Program on AIDS / Thai Red Cross Society, Bangkok, Thailand
- Policlinica Metropolitana, Caracas, Venezuela